CLINICAL TRIAL: NCT07261176
Title: Effect of Smoking on Retinal Vessel Morphology and Functionality: A Case-Control, Clinical Trial
Brief Title: Effect of Smoking on Retinal Vessel Morphology and Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Querques Giuseppe, Associate Professor, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SMOKE-DVA
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Smokers
Keywords: smoke

STUDY DESIGN:
Intervention Model Description: Case-control design with two parallel groups: smokers receiving intervention (smoking one cigarette) and non-smoking controls undergoing examinations at matched time intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers Group (Experimental): Twenty healthy volunteers with regular daily tobacco activity (approximately 10 cigarettes per day, smoking duration 5-10 years, using cigarettes with 0.8 grams nicotine content). Participants underwent OCT-A, DVA, and RVA examinations at baseline, 3 minutes, and 30 minutes after smoking one cigarette.
  Interventions: Behavioral: Cigarette Smoking
- Non-smokers Control Group (No Intervention): Twenty healthy volunteers with no tobacco activity as normal life habit. Control participants underwent the same OCT-A, DVA, and RVA examinations at baseline, 8 minutes, and 35 minutes (corresponding timepoints without smoking) to assess examination variability and learning effects.

INTERVENTIONS:
Behavioral: Cigarette Smoking — Participants smoked one cigarette containing 0.8 grams of nicotine under standardized conditions. Participants were required to abstain from tobacco activity for 24 hours prior to baseline examination and to avoid vasoconstrictor substances (coffee, alcohol) before examinations.
  Arms: Smokers Group

SUMMARY:
The study aims at evaluating the effect of smoking activity on anatomy and functionality of retinal blood vessels using optical coherence tomography angiography (OCT-A) and dynamic vessel analysis (DVA).

This is a low-risk, single-center, case-control, interventional clinical trial. Forty healthy subjects were enrolled: 20 healthy volunteers with regular daily tobacco activity (approximately 10 cigarettes per day for 5-10 years) and 20 healthy volunteers with no tobacco activity as controls.

Each subject underwent comprehensive ophthalmologic examination including OCT-A, DVA, and retinal vessel analysis (RVA) at baseline. Examinations were repeated for the smoking group at 3 and 30 minutes after smoking activity, and for controls at 8 and 35 minutes after baseline to assess examination variability.

The primary outcomes assessed changes in retinal perfusion and retinal vascular response after cigarette smoking compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes (age 20 to 30 years old)
* Healthy volunteers who can understand and sign informed consent
* For Smokers Group: Regular daily tobacco activity (approximately 10 cigarettes per day, smoking duration 5-10 years, using cigarettes with 0.8 grams nicotine content)
* For Control Group: No tobacco activity as normal life habit
* Willing to abstain from tobacco activity for 24 hours prior to baseline examination
* Willing to avoid vasoconstrictor substances (coffee, alcohol) prior to examinations

Exclusion Criteria:

* Inability to follow planned procedures
* Opacity of dioptric media (lens, cornea, or vitreous) that prevents execution of examinations
* Known allergies that do not allow pupillary dilation
* Ocular pathologies
* Systemic hypertension
* Diabetes mellitus
* Myopia greater than -8.0 Diopters (D)
* Hyperopia greater than +5.0 D
* Astigmatism greater than -3.0 D

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Central Retinal Artery Equivalent (CRAE) | Baseline, 3 minutes and 30 minutes post-smoking (smokers); baseline, 8 minutes and 35 minutes (controls)
  Changes in central retinal artery equivalent measured using Retinal Vessel Analyzer (RVA). CRAE relates to the diameter of the central retinal artery, expressed in measurement units (MU). Higher values indicate larger arterial diameter.
Arterial Dilation Percentage Post-Flicker Stimulation | Baseline, 3 minutes and 30 minutes post-smoking (smokers); baseline, 8 minutes and 35 minutes (controls)
  Percentage increase in retinal arterial vessel diameter in response to flicker light stimulation measured by Dynamic Vessel Analyzer (DVA). Calculated as percentage increase in vessel diameter relative to baseline after 20 seconds of flicker stimulation, averaged across 3 measurement cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandello, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Università Vita Salute San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu X, Yang K, Xiao Y, Ye C, Zheng J, Su B, Zheng Y, Zhang X, Shi K, Li C, Lu F, Qu J, Li M, Cui L. Association of cigarette smoking with retinal capillary plexus: an optical coherence tomography angiography study. Acta Ophthalmol. 2022 Nov;100(7):e1479-e1488. doi: 10.1111/aos.15157. Epub 2022 Apr 9. PMID 35396902
- [Background] Garhofer G, Resch H, Sacu S, Weigert G, Schmidl D, Lasta M, Schmetterer L. Effect of regular smoking on flicker induced retinal vasodilatation in healthy subjects. Microvasc Res. 2011 Nov;82(3):351-5. doi: 10.1016/j.mvr.2011.07.001. Epub 2011 Jul 12. PMID 21771603
- [Background] Ciesielski M, Rakowicz P, Stopa M. Immediate effects of smoking on optic nerve and macular perfusion measured by optical coherence tomography angiography. Sci Rep. 2019 Jul 15;9(1):10161. doi: 10.1038/s41598-019-46746-z. PMID 31308472
- [Background] Siedlecki J, Mohr N, Luft N, Schworm B, Keidel L, Priglinger SG. Effects of Flavanol-Rich Dark Chocolate on Visual Function and Retinal Perfusion Measured With Optical Coherence Tomography Angiography: A Randomized Clinical Trial. JAMA Ophthalmol. 2019 Dec 1;137(12):1373-1379. doi: 10.1001/jamaophthalmol.2019.3731. PMID 31556937
- [Background] McClintic SM, Jia Y, Huang D, Bailey ST. Optical coherence tomographic angiography of choroidal neovascularization associated with central serous chorioretinopathy. JAMA Ophthalmol. 2015 Oct;133(10):1212-4. doi: 10.1001/jamaophthalmol.2015.2126. No abstract available. PMID 26135638
- [Background] Huang Y, Zhang Q, Thorell MR, An L, Durbin MK, Laron M, Sharma U, Gregori G, Rosenfeld PJ, Wang RK. Swept-source OCT angiography of the retinal vasculature using intensity differentiation-based optical microangiography algorithms. Ophthalmic Surg Lasers Imaging Retina. 2014 Sep-Oct;45(5):382-9. doi: 10.3928/23258160-20140909-08. PMID 25230403
- [Background] de Carlo TE, Romano A, Waheed NK, Duker JS. A review of optical coherence tomography angiography (OCTA). Int J Retina Vitreous. 2015 Apr 15;1:5. doi: 10.1186/s40942-015-0005-8. eCollection 2015. PMID 27847598
- See also: IRCCS Ospedale San Raffaele Official Website — https://www.hsr.it
- See also: Vita-Salute San Raffaele University — https://www.unisr.it